CLINICAL TRIAL: NCT04895852
Title: Efficacy and Safety of Transcutaneous Electrical Acupoints Stimulation for Preoperative Anxiety in Thoracoscopic Surgery: Study Protocol for a Randomized Controlled Trial
Brief Title: Clinical Study of TEAS Intervention in Relieving Anxiety Before Thoracoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20210427
Record Dates: First submitted 2021-04-27; First posted 2021-05-20 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Acupuncture Therapy; Preoperative Period; Anxiety; Thoracoscopic Surgery
Keywords: Acupuncture Treatment; Preoperative Conditioning; Anxiety; Thoracoscopic Surgery
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAS group (Experimental): 30 minutes TEAS therapy on DU20, EX-HN3, LI4, LR3 once per day for three days before surgery.
  Interventions: Device: TEAS
- Control group (Sham Comparator): The control group selects the same acupoints as the TEAS group and other intervention measures are the same as the TEAS group except for the current intensity is set to 0-mA.
  Interventions: Device: Sham TEAS

INTERVENTIONS:
Device: TEAS — The self-adhesive gel electrode pad will be placed at the center of DU20 (Baihui), EX-HN3 (Yintang) and both sides of LI4 (Hegu), LR3 (Taichong) in strict accordance with the World Health Organization Standardized Acupuncture Location. Electric stimulation will be used with a TEAS apparatus (HANS200A Beijing Huawei Co., LTD.) . The frequency of the electrical stimulation will be set as alternating 2/100Hz to relieve anxiety. The current intensity will be adjusted individually, starting at 1 mA and increasing gradually until the patient can perceive and tolerate it (preferably slight twitching of local muscles without pain).
  Arms: TEAS group
Device: Sham TEAS — The STEAS group selects the same acupoints as the TEAS group and other intervention measures are the same as the TEAS group except for the current intensity is set to 0-mA. The acupuncturist responsible for the operation will tell patients in STEAS group that this is a type of stimulus without perception.
  Arms: Control group

SUMMARY:
This single-center randomized sham-controlled trial will be conducted in cardiothoracic surgery department of the Yueyang Hospital of Integrated Traditional Chinese and Western Medicine in China. A total of 92 eligible participants with pulmonary nodules (size ≥ 8mm) who will undergo VATS will be randomly allocated to a TEAS group and a sham TEAS (STEAS) group in a 1:1 ratio. Daily TEAS/STEAS treatment will be performed starting on 3 days before the VATS and continued for three consecutive days, once per day. The primary outcome will be the minimal clinically important difference of generalized anxiety disorder scale score change between the day before surgery with the baseline. The secondary outcomes include serum concentrations of 5-hydroxytryptamine, norepinephrine and gamma-aminobutyric acid, intraoperative anesthetic consumption, time to postoperative chest tube removal, postoperative pain, length of postoperative hospital stay. The adverse events will be recorded for safety evaluation. All data in the study will be analyzed using the SPSS 21.0 statistical software package.

DETAILED DESCRIPTION:
This single center, randomized, sham-controlled, participant-blinded and assessor-blinded trial will be conducted at the inpatient ward of cardiothoracic surgery department of Yueyang Hospital of Integrated Traditional Chinese and Western Medicine affiliated to Shanghai University of Traditional Chinese Medicine. The trial will commence after ethical approval has been obtained and the protocol has been registered. Patient enrollment started in late June 2021 and is expected to end in March 2023. An estimated 92 participants will be recruited and randomly assigned to receive TEAS or sham TEAS (STEAS) in a l:l ratio using SPSS 21.0 software. During the development of the standard protocol, the Standards for Reporting Interventions in Clinical Trials for Acupuncture (STRICTA) and the SPIRIT reporting guidelines will be followed to explicitly and transparently explain the therapeutic processes involved.

Patients who will undergo VATS for pulmonary nodules will be screened. . Potential subjects will be interviewed preoperatively by the clinical research coordinator to assess whether they meet the inclusion and exclusion criteria. Eligible participants will voluntarily provide written informed consent prior to randomization.

This study will have a single-blind design. The patients are blinded to the group assignment and are told that they might or might not feel a sensation when the TEAS is working. Both acupoint stimulations in the TEAS group and in the STEAS group will be performed by the same acupuncturist who is not involved in the process of data collection. The TEAS instrument is covered with an opaque box for adequate blinding. The randomized numbers were generated with SPSS 21.0 (IBM®SPSS®Statistics, Version 21) software. The random sequence for group classification will be sealed in a confidential envelope. Patients will be randomly allocated into the TEAS group or STEAS group at a ratio of 1:1. Group assignment was exposed from a sealed envelope only by an acupuncturist. Patients will be treated separately to prevent communication. Efficacy evaluation will be conducted blinded to the grouping allocation. The efficacy evaluators and statisticians will be separated and blinded. To test the participant-blinding effects, all participants will be asked to guess whether they had received TEAS or STEAS within 5 minutes after one of the treatment sessions before VATS.

ELIGIBILITY:
Inclusion criteria

1. Those diagnosed as pulmonary nodules requiring VATS.
2. Age between 18 and 75 years old.
3. 4 ≤ GAD-7 score ≤ 9 and those who have no previous mental illness and have not used anti-anxiety or psychotropic drugs within 2 weeks.
4. Those who have clear consciousness, normal understanding, no expression barriers, can cooperate with treatment and have signed an informed consent.
5. Patients who have not received TEAS treatment in the past.
6. Patients who have not participated or participating in other clinical trials one month before enrollment.

Exclusion criteria

1. Patients with skin infections in local meridian points.
2. Patients with upper or lower limb nerve injury.
3. Patients who had been implanted pacemaker.

Rejection, suspension and dropout criteria

1. Those with serious adverse reactions.
2. Those who presented worsen symptoms or life-threatening illnesses that cannot be continued during treatment.
3. The principal investigator asserts that there are unacceptable risks for serious adverse events during the study.
4. Patients who cannot cooperate to complete the research plan, including language difficulties, infectious diseases and other medical history.
5. Patients quit by themselves.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-01-11 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Score change of Generalized Anxiety Scale (GAD-7) | up to 3 days before surgery
  Add the scores of each of the 7 items to get the total score; among them, 0-4 points for no anxiety, 5-9 points for possible mild anxiety, 10-14 points for possible moderate anxiety, 15 Scores above are likely to have severe anxiety. The GAD-7 scores' Change between three days before and the day before surgery will be recorded.

SECONDARY OUTCOMES:
5-HT（µmol/L） | on the third day before the treatment and the day before the operation
  The blood of each group of patients was collected on the third day before the treatment and the day before the operation, and the levels of neurotransmitter indexes (5-HT, NE, GABA) in the peripheral blood were detected by the immunoturbidimetric method.
NE（µg/L） | on the third day before the treatment and the day before the operation
  The blood of each group of patients was collected on the third day before the treatment and the day before the operation, and the levels of neurotransmitter indexes (5-HT, NE, GABA) in the peripheral blood were detected by the immunoturbidimetric method.
GABA（µmol/L） | on the third day before the treatment and the day before the operation
  The blood of each group of patients was collected on the third day before the treatment and the day before the operation, and the levels of neurotransmitter indexes (5-HT, NE, GABA) in the peripheral blood were detected by the immunoturbidimetric method.
Chest tube removal time | up to 168 hours after surgery
  Record the time from the end of surgery to the removal of chest tube.
Postoperative pain | up to 2 days after surgery
  VAS ranges from 0 (no pain) to 10 (unbearable pain). A change of 10 for the 100mm pain VAS signify a clinically important improvement or deterioration. Participants will be asked to describe their average surgical incision intensity in the 48 hours after surgery.
Length of postoperative hospital stay | up to 14 days after surgery
  The length of postoperative stay will be recorded.
Intraoperative anesthetic consumption | From the beginning to the end of the surgery
  The types and cumulative doses of intraoperative analgesics will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Zhou, Study Director — Yueyang Hospital of Integrated Traditional Chinese and Western Medicine
Locations (1):
- Shanghai Yueyang Integrated Medicine Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Reasonable requests for IPD data can be obtained by contacting the investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within five years of publication of the trial.
Access Criteria: Reasonable requests for IPD data can be obtained by contacting the investigator.

REFERENCES:
- [Derived] Wu X, Chen T, Wang K, Wei X, Feng J, Zhou J. Efficacy and safety of transcutaneous electrical acupoints stimulation for preoperative anxiety in thoracoscopic surgery: study protocol for a randomised controlled trial. BMJ Open. 2023 Feb 16;13(2):e067082. doi: 10.1136/bmjopen-2022-067082. PMID 36797022